CLINICAL TRIAL: NCT04104503
Title: Interventional, Open-label, Two-part, Partly-randomized Study Investigating the Pharmacokinetic Properties, Absolute Bioavailability, Food Effect, and Intra-subject Variability of up to 5 Prototype Modified-release Tablet Formulations of Lu AF11167 in Healthy Subjects
Brief Title: A Study Investigating Tablet Formulations of Lu AF11167 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18153A
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental)
  Interventions: Drug: Lu AF11167
- Part B group 1 (Experimental): Treatment period 1: Fasted + iv;
  Treatment period 2: Fasted;
  Treatment period 3: High-fat meal
  Interventions: Drug: [14C]-Lu AF11167; Drug: Lu AF11167 MR tablet prototype formulation selected from part A or 1 mg modified release tablet (reference formulation)
- Part B group 2 (Experimental): Treatment period 1: High-fat meal;
  Treatment period 2: Fasted + iv;
  Treatment period 3: Fasted
  Interventions: Drug: [14C]-Lu AF11167; Drug: Lu AF11167 MR tablet prototype formulation selected from part A or 1 mg modified release tablet (reference formulation)
- Part B group 3 (Experimental): Treatment period 1: Fasted;
  Treatment period 2: High-fat meal;
  Treatment period 3: Fasted + iv
  Interventions: Drug: [14C]-Lu AF11167; Drug: Lu AF11167 MR tablet prototype formulation selected from part A or 1 mg modified release tablet (reference formulation)

INTERVENTIONS:
Drug: Lu AF11167 — Lu AF11167 - 2 mg modified release tablets (reference formulation), up to 5 prototype MR tablet formulations (test formulations)
  Arms: Part A
Drug: [14C]-Lu AF11167 — single iv microdose administered as a 15 minutes infusion
  Arms: Part B group 1; Part B group 2; Part B group 3
Drug: Lu AF11167 MR tablet prototype formulation selected from part A or 1 mg modified release tablet (reference formulation) — Single oral dose
  Arms: Part B group 1; Part B group 2; Part B group 3

SUMMARY:
The purpose of this study is to investigate the extent to which Lu AF11167 enters the bloodstream following tablet intake and the influence of food on uptake in healthy men and women

DETAILED DESCRIPTION:
This study will be split into Part A and Part B. Part A will happen first and will look at new tablet formulations of the test medicine compared to a previously known formulation (reference tablet). The results from Part A of the study will be used to decide which formulation will be tested in Part B of the study. Part B of the study will look at the food effect, variability between participants, and absolute bioavailability of the test medicine i.e. how much of the test medicine is taken up by the body when dosed by mouth compared to when dosed once by injection directly into the vein. Safety and tolerability will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of ≥18.5 and ≤30.0 kg/m2
* (Part B only) Women of child-bearing potential will have a confirmed non-pregnant and non-lactating status

Exclusion Criteria:

* The subject has any concurrent disorder that may affect the particular target or absorption, distribution, or elimination of the investigational medical product

Other in- and exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Cmax of Lu AF11167 | From 0 to 48 hours
  Maximum observed plasma concentration
AUC(0-inf) of Lu AF11167 | From 0 to 48 hours
  Area under the plasma concentration time curve from zero to infinity
Relative bioavailability F(rel) of Lu AF11167 | From 0 to 48 hours
  F(rel) is estimated as the dose normalized AUC(inf) for the test formulation relative to the reference formulation (part A only)
Absolute bioavailability F(abs) of Lu AF11167 | From 0 to 48 hours
  F(abs) is estimated as the dose normalized AUC(inf) for the test formulation relative to the intravenous reference formulation (part B only)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Quotient, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided